CLINICAL TRIAL: NCT00269815
Title: Long-term Safety and Effectiveness of OROS (Methylphenidate HCl) in Children With ADHD
Brief Title: Long-term Safety and Effectiveness of OROS Methylphenidate HCl in Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR006001
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; OROS®; children; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

ARMS (1):
- 001 (Experimental): methylphenidate HCl
  Interventions: Drug: methylphenidate HCl

INTERVENTIONS:
Drug: methylphenidate HCl

SUMMARY:
The purpose of this study is to evaluate the long-term safety and effectiveness of OROSÂ® Methylphenidate HCl (a central nervous system stimulant) in children with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) represents the most common neurobehavioral disorder in children, affecting 3% to 5% of the school-age population. Behavioral pediatricians, child psychiatrists, and child neurologists indicate that referrals for ADHD may constitute up to 50% of their practices. This is a multicenter, open-label, non-randomized, single-treatment study in children 6 to 13 years of age with ADHD who have successfully completed specific earlier ALZA studies. Part I of this study will evaluate the safety and effectiveness of OROS® (methylphenidate HCl) for a period of one year in children with ADHD. Part II of this study continues the evaluation of the safety and effectiveness of OROS® (methylphenidate HCl) in children with ADHD who have completed one year in Part I of the study. During Part I of the study, patients will be assigned to treatment with OROS® (methylphenidate HCl) 18, 36, or 54 milligrams once daily, as determined by the results from their participation in earlier ALZA studies. Patients continuing in Part II of the study continue to receive a daily dose as determined from the dosing at the end of Part I. Doses can be titrated up or down, as considered appropriate by the medical personnel at the study site, with a maximum once-daily dose of 54 milligrams. Effectiveness is determined by standardized measurements of attention, behavior, and hyperactivity including: the IOWA (Inattention Overactivity with Aggression) Conners Rating Scale, Inattention/Overactivity (I/O) and Oppositional/Defiance (O/D) subscales; Peer Interaction assessment; Global evaluation of effectiveness of therapy; and the Parent Satisfaction Questionnaire. Safety evaluations include the incidence of adverse events, physical examinations, clinical laboratory tests, vital signs, sleep quality, appetite, and the presence/severity of tics (hard-to-control, repeated twitching of any parts of the body or hard-to-control repeating of sounds or words).

Data will be summarized and no formal hypotheses will be tested. Part I: A daily morning oral dose of 18, 36, or 54 milligrams of OROS® (methylphenidate HCl) for up to 12 months. Part II: Continuation for up to 15 months of the same daily dose taken at the end of Part I. Total treatment duration to approximately 27 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have successfully completed one of the following earlier ALZA studies: CR005992, C-97-033 (and then successfully completed C-98-011), CR005989, or CR005995, without significant drug-related adverse events
* whose primary care physician agrees that it is appropriate to participate in this study
* who agree to take only the OROS® (methylphenidate HCl) supplied and no other methylphenidate dosage form or other medications for the treatment of ADHD during the study
* who are able to comply with the study visit schedule and whose parent(s) and teachers are willing and able to complete the protocol-specified assessments
* who have normal urinalysis, hematological and blood chemistry values or, if values are outside the normal range, they are determined not clinically significant by the investigator

Exclusion Criteria:

* Patients having clinically significant gastrointestinal problems, including narrowing of the gastrointestinal tract
* having any coexisting medical condition or are taking any medication that is likely to interfere with safe administration of methylphenidate
* having a known hypersensitivity to methylphenidate
* having a history of high blood pressure or who have a blood pressure (systolic or diastolic) equal to or greater than the 95th percentile for age, gender and height
* if female, have begun menstruation

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events; Changes in physical examinations, clinical laboratory tests, vital signs, sleep quality, appetite, and tics

SECONDARY OUTCOMES:
IOWA (Inattention Overactivity with Aggression) Conners Rating Scale, Inattention/Overactivity (I/O) and Oppositional/Defiance (O/D) subscales; Peer Interaction assessment; Global evaluation of effectiveness of therapy; Parent Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Result] Wilens T, McBurnett K, Stein M, Lerner M, Spencer T, Wolraich M. ADHD treatment with once-daily OROS methylphenidate: final results from a long-term open-label study. J Am Acad Child Adolesc Psychiatry. 2005 Oct;44(10):1015-23. doi: 10.1097/01.chi.0000173291.28688.e7. PMID 16175106